CLINICAL TRIAL: NCT06420986
Title: Open Hemorrohoidectomy Versus Transanal Hemorrhoidal Desarterialization in Hemorrhoids Grade III: The Effect on Symptons: An Open-label Randomized Controlled Trial
Brief Title: Open Hemorrohoidectomy Vs Transanal Hemorrhoidal Desarterialization in Hemorrhoids Grade III: The Effect on Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Son Llatzer (Other)
Collaborators: Fundació d'investigació Sanitària de les Illes Balears (Other Government)
Responsible Party: Principal Investigator, Ignacio Fernandez Hurtado, Specialist in General Surgery. Specialist in Digestive Surgery, Hospital Son Llatzer
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IB4323-20PI
Record Dates: First submitted 2024-05-15; First posted 2024-05-20 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Hemorrhoids Third Degree
Keywords: hemorrhoids third degree; botulinum Toxin; Hemorrhoidectomy; Transanal Hemorrhoidal Dearterialization; hemorrhoidal Disease Symptom Score

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hemorrhoidectomy (Experimental)
  Interventions: Procedure: Open Hemorrhoidectomy
- Transanal Hemorrhoidal Dearterialization (Experimental)
  Interventions: Procedure: Transanal Hemorrhoidal Dearterialization

INTERVENTIONS:
Procedure: Open Hemorrhoidectomy — Surgical treatment of Hemorrhoids. Removal of hemorrohids leaving the wounds open. Surgical technique described by Milligan Morgan
  Arms: Hemorrhoidectomy
Procedure: Transanal Hemorrhoidal Dearterialization — Surgical treatment of Hemorrhoids. This operation involves no excision. The hemorrhoidal arteries are ligated and the hemorrhoial prolapse is treated by a suture mucopexi. Described by Rato
  Arms: Transanal Hemorrhoidal Dearterialization

SUMMARY:
The goal of this clinical trial is to learn if open hemorroidectomy diminishes symptoms compared to transanal hemorrhoidal desarterialization (THD) in patients presenting with hemorrhoids grade III. The main question it aims to answer is:

- Do patients undergoing open hemorroidectomy present with lesser symptoms 1 year after surgery, compared to those undergoing a THD?

Researchers will compare open hemorroidectomy to THD in terms of symptom response one year after the procedure.

Participants will:

* Undergo surgical treatment of hemorroids performed by one of the two techniques: open hemorroidectomy versus THD.
* Fill in symptom forms before and one year after the surgical procedure.
* Attend control visits one week, one month, three months and one year after the surgical procedure.

ELIGIBILITY:
Inclusion criteria:

* Age older than 18.
* Hemorroids grade III.
* Surgical indication for hemorroid treatment.
* Signed informed consent.

Exclusion criteria:

* Acute hemorroidal disease.
* Previous hemorroidal surgery.
* Concomitant anal fissure.
* Concomitant perianal fistulae.
* Concomitant rectal prolapse.
* Inflamatory bowel disease.
* Anal or colorrectal cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2024-04-17 (Actual)

PRIMARY OUTCOMES:
hemorrhoidal disease symptom score | one year
  A score that defines the frecuency of pain, pruritus, bleeding, soiling and prolapse. Score 0 to 20. Higher scores mean a worse outcome
short health scale in hemorrhoidal disease | one year
  a subjective scale which defines symptom intensity, the patient's worrying and the role in impairment of daily activity. Score 4 to 28. Higher scores mean a worse outcome

SECONDARY OUTCOMES:
postoperative pain | 1 week after surgical procedure
  pain measured in visual analogic scale (VAS) Scale: 0 to 10. Higher scores mean a worse outcome
fecal incontinence | baseline and 1 week, 3 months and 1 year after surgical procedure
  measured in Wexner scale. Score 0 to 20. Higher scores mean a worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Son Llatzer, Palma de Mallorca, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fernandez-Hurtado I, Pages-Valle N, Sarubbo MF, Claramonte-Bellmunt O, Baena-Bradaschia S, Cifuentes-Rodenas JA, Serra-Aracil X. Open excisional haemorrhoidectomy versus transanal haemorrhoidal dearterialization for grade III haemorrhoids: open-label randomized clinical trial. Br J Surg. 2025 Dec 24;113(1):znaf282. doi: 10.1093/bjs/znaf282. PMID 41553737